CLINICAL TRIAL: NCT04011748
Title: Clinical Treatment of Alopecia Areata With Stem Cell Educator Therapy
Brief Title: Clinical Application of Stem Cell Educator Therapy in Alopecia Areata
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Throne Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-TH-001
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis

STUDY DESIGN:
Intervention Model Description: AA subjects will receive the treatment with Stem Cell Educator therapy
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Hair regrowth by SCE (Experimental): AA subjects will receive Stem Cell Educator therapy. Hair regrowth will be evaluated during six-month follow-up studies.
  Interventions: Combination Product: Stem Cell Educator therapy
- Minoxidil therapy (Experimental): Control subjects will receive treatment with topical 5% minoxidil
  Interventions: Combination Product: Stem Cell Educator therapy

INTERVENTIONS:
Combination Product: Stem Cell Educator therapy — AA subjects will be recruited and followed by the treatment with SCE therapy.

SUMMARY:
Alopecia areata (AA) is a common autoimmune disease that results in loss of body hair in varying degrees. The condition is estimated to affect more than 6.8 million people in the United States alone (naaf.org), with a worldwide prevalence of 0.1% to 0.2% and calculated lifetime risk of 2%. AA is the most common form of the disease, in which areas of complete hair loss arise within normal hair-bearing skin. Other forms include alopecia totalis (AT), characterized by total loss of scalp hair, and alopecia universalis (AU), characterized by complete loss of body hair. AA and its variants can have devastating effects on patients' quality of life and social functioning. At present, curative therapy for AA does not exist. Therapeutic options are currently very limited, such as intralesional injections of glucocorticoids and induction of allergic contact dermatitis. These therapies are not effective for many patients and are generally impractical for patients with diffuse AA, AT or AU. Recently, Janus kinase (JAK) inhibitors were effective for the treatment of severe AA. However, for those patients who do respond, relapses are common after discontinuation of treatment, due to the existing of autoimmune memory T cells. Stem Cell Educator (SCE) therapy, which uses only autologous mononuclear cells that are externally exposed to cord blood stem cells, has previously been proven safe and effective in subjects for the improvement of type 1 diabetes (T1D), T2D and other autoimmune diseases such as alopecia areata. Minoxidil is the FDA approved drug for the treatment of androgenetic alopecia (AGA) in 1988. This trial will explore the therapeutic potential of Stem Cell Educator therapy for the treatment of AA by using topical minoxidil as control.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ( 18 years)
2. Must have a clinical diagnosis of AA, at least 50% hair loss involving the scalp
3. For cases in which there is 80% or more scalp hair loss, the duration of the severity of hair loss must be 10 years or less
4. Stable or worsening hair loss for at least 6 months without evidence of hair regrowth
5. Patients must not have received any treatments known to affect AA within 2 months of screening
6. Patients must agree that they are not permitted to use any other treatment besides topical minoxidil known to affect AA during a period of 6 months after undergoing SCE therapy
7. Adequate venous access for apheresis
8. Ability to provide informed consent
9. For female patients only, willingness to use FDA-recommended birth control (http://www.fda.gov/downloads/ForConsumers/ByAudience/ForWomen/FreePublications/UCM356451.pdf) until 6 months post treatment.
10. Must agree to comply with all study requirements and be willing to complete all study visits

Exclusion Criteria:

1. AST or ALT 2 > x upper limit of normal.
2. Abnormal bilirubin (total bilirubin > 1.2 mg/dL, direct bilirubin > 0.4 mg/dL)
3. Creatinine > 2.0 mg/dl.
4. Known coronary artery disease or EKG suggestive of coronary artery disease unless cardiac clearance for apheresis is obtained from a cardiologist.
5. Known active infection such as Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV)
6. Pregnancy assessed by a positive serum pregnancy test or breastfeeding mothers
7. Use of immunosuppressive medication within one month of enrollment including but not limited to prednisone, cyclosporine, tacrolimus, sirolimus, and chemotherapy.
8. Presence of any other autoimmune diseases (lupus, rheumatoid arthritis, scleroderma, etc.)
9. Anticoagulation other than ASA.
10. Hemoglobin < 10 g/dl or platelets < 100 k/ml
11. Is unable or unwilling to provide informed consent
12. Presence of any other physical or psychological medical condition that, in the opinion of the investigator, would preclude participation
13. Significant cardiovascular diseases that would make use of oral minoxidil inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
The percentage change in scalp hair growth. | Hair regrowth will be evaluated at different time points post receiving Stem Cell Educator therapy in 1, 3, and 6 months.
  The primary endpoint was the percentage change in scalp hair growth, measured with the Severity of Alopecia Tool (SALT) score.

SECONDARY OUTCOMES:
Feasibility of SCE therapy | 6 months
  The feasibility will be determined by the number of patients who were unable to complete SCE Therapy.
Preliminary efficacy of SCE therapy | 6 months
  This will be determined by the duration of maintaining hair growth following SCE therapy.
Efficacy of modulation of autoimmune-related memory T-cell markers | 6 months
  Measurements of immune markers' changes will be preformed by flow cytometry such as CD8+CD45RO+CCR7- effector memory T cells. Peripheral blood mononuclear cells (PBMC) will be collected at 1, 3, 6 month post the SCE therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Throne Biotechnologies, Paramus, New Jersey, United States

REFERENCES:
- [Background] Zhao Y, Knight CM, Jiang Z, Delgado E, Van Hoven AM, Ghanny S, Zhou Z, Zhou H, Yu H, Hu W, Li H, Li X, Perez-Basterrechea M, Zhao L, Zhao Y, Giangola J, Weinberg R, Mazzone T. Stem Cell Educator therapy in type 1 diabetes: From the bench to clinical trials. Autoimmun Rev. 2022 May;21(5):103058. doi: 10.1016/j.autrev.2022.103058. Epub 2022 Jan 31. PMID 35108619
- [Result] Li Y, Yan B, Wang H, Li H, Li Q, Zhao D, Chen Y, Zhang Y, Li W, Zhang J, Wang S, Shen J, Li Y, Guindi E, Zhao Y. Hair regrowth in alopecia areata patients following Stem Cell Educator therapy. BMC Med. 2015 Apr 20;13:87. doi: 10.1186/s12916-015-0331-6. PMID 25896390
- [Result] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Yin Z, Li H, Zhang Y, Diao Y, Li Y, Chen Y, Sun X, Fisk MB, Skidgel R, Holterman M, Prabhakar B, Mazzone T. Reversal of type 1 diabetes via islet beta cell regeneration following immune modulation by cord blood-derived multipotent stem cells. BMC Med. 2012 Jan 10;10:3. doi: 10.1186/1741-7015-10-3. PMID 22233865
- [Result] Zhao Y. Stem cell educator therapy and induction of immune balance. Curr Diab Rep. 2012 Oct;12(5):517-23. doi: 10.1007/s11892-012-0308-1. PMID 22833322
- See also: Throne Biotechnologies Inc — https://thronebio.com/